CLINICAL TRIAL: NCT00879723
Title: Burn Micronutrient Repletion Pilot Study: Characterizing Relationships Between Vitamin and Mineral Supplementation and Health Outcomes of Adult Burn Patients
Brief Title: Burn Micronutrient Repletion Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Collaborators: Memorial Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-SIUSOM-09-002-1; SCRIHS 08-105
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Burn
Keywords: post-burn recovery; oxidative stress; micronutrient protocol
MeSH Terms: conditions — Burns | interventions — Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin and mineral supplementation (Experimental): Intravenous micronutrient solution or an oral micronutrient supplementation twice per day for 14 days. Treatment is determined by percent total body surface area burned.
  Interventions: Dietary Supplement: Vitamin and Mineral supplementation
- Control (No Intervention): current vitamin regimen as listed on the Memorial medical Center Order Set for burn unit admission.

INTERVENTIONS:
Dietary Supplement: Vitamin and Mineral supplementation — IV - 2x per day given 2 - 12 hours apart. A.M. solution - Infuvite multivitamin with minerals, Selenium 200mcg, Zinc 30mg, Vitamin B1 100mg and Vitamin C 500mg. P.M. solution - Cuperic Chloride 9mg (provides Copper 3.36mg) and Vitamin C 500mg. Each fluid solution will run for 4 hours.
  Enteral (oral) 2 x per day given 2 - 12 hours apart. A.M. dose - multivitamin with minerals, Selenium 200mcg, Zinc 30mg, Vitamin B1 100mg and Vitamin C 500mg. P.M. dose - Copper 4mg and Vitamin C 500mg.
  Arms: Vitamin and mineral supplementation

SUMMARY:
Burn injury patients undergo a series of metabolic changes that, if untreated, could lead to reduced health outcomes. Nutrition is thought to play a vital role in post-burn recovery. The research team developed a novel vitamin and mineral supplementation protocol based on current scientific literature. The study will test the hypothesis that the novel vitamin and mineral supplement regimen will improve adult patient recovery from burn injury.

DETAILED DESCRIPTION:
Burn injury patients undergo a series of metabolic events that, if untreated, could lead to severe physical impairment and even death. Antioxidants minimize free radical damage by neutralizing the chemical reaction as well as promoting cellular repair. Currently there is no consistent protocol for micronutrient repletion in adult burn patients. The aim of this study is to evaluate the effectiveness of the current vitamin regimen in comparison to the novel vitamin and mineral supplementation protocol developed by the research team. Dosages for oral and intravenous supplementation are based on current literature. The combination of intravenous and enteral treatment is important due to gastrointestinal mucosal swelling related to post-burn fluid resuscitation. Measurable health outcomes will include rate of infection, length of hospital stay, mortality rate, hospital cost, number of days in intensive care unit, number of ventilator-dependent days and wound healing. The investigators hypothesize that use of the novel vitamin and mineral supplement regimen will improve adult burn patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients who present at the burn unit with TBSA > 1%

Exclusion Criteria:

* less than 19 years old
* chronic renal failure
* chronic liver failure
* pregnancy or lactation
* patients who require parenteral nutrition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
wound healing | 14 days

SECONDARY OUTCOMES:
rate of infection | 14 days
number of days in hospital | 14 days
number of days in Intensive Care Unit | 14 days
number of days on ventilator | 14 days
mortality rate | 14 days
hospital charges | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Neumeister, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Memorial Medical Center, Springfield, Illinois, United States